CLINICAL TRIAL: NCT01942226
Title: Investigation on Medical Management of Dry Eye Patients
Status: Completed | Type: Observational
Sponsor: National Cheng Kung University (Other)
Collaborators: National Taiwan University Hospital (Other); Sun-Huei Tseng Eye Institute (Unknown); Institute of Clinical Pharmacy and Pharmaceutical Sciences, National Cheng Kung University, Tainan, Taiwan (Unknown); Allergan Pharmaceuticals Taiwan Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yea-Huei Kao Yang, Professor, National Cheng Kung University
Other Study IDs: MODE
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Dry eye is a common complaint in patients encountered by ophthalmologists, which may result from the inflammatory response and can occur in the absence of systemic disease. However, the management of dry eye syndrome in real setting warrants assessment but remains lacking in Taiwan. We conducted an perspective observational study to evaluate the medical management of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Have given a written informed consent
* Clinical diagnosis of dry eye syndrome
* Have at least one Schirmer's test positive result (less than 10mm/5min) in at least one eye within one year

Exclusion Criteria:

* Pregnancy
* Cognitive or psychiatric deficit that precludes informed consent
* Cognitive or psychiatric deficit that precludes ability to perform requirements of the investigation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from a primary care clinic or a tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Artificial tears utilization patterns | within 1 month before recruitment

SECONDARY OUTCOMES:
Changes of dry eye symptoms, evaluated by clinicians | Baseline
  Measured by clinical global impression (CGI)
Changes of dry eye symptoms, evaluated by patients | Baseline
  Measured by subject global assessment (SGA)

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Huei Kao Yang, Professor, Principal Investigator — Institute of Clinical Pharmacy and Pharmaceutical Sciences, National Cheng Kung University
Locations (2):
- Taiwan (2):
  - Sun-Huei Tseng Eye Institute, Tainan
  - Department of Ophthalmology, National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Yeh PT, Chien HC, Ng K, Tseng SH, Chen WL, Hou YC, Wang IJ, Chu HS, Kao Yang YH, Hu FR. Concordance between patient and clinician assessment of dry eye severity and treatment response in Taiwan. Cornea. 2015 May;34(5):500-5. doi: 10.1097/ICO.0000000000000409. PMID 25782401